CLINICAL TRIAL: NCT05860387
Title: Early Diagnosis of Invasive Lung Aspergillosis
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: Public Health Institute Ostrava (Unknown); University Hospital Olomouc (Other); Municipal Hospital Ostrava (Other); Havířov Hospital (Unknown); Krnov Hospital (Unknown); University of Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: EDILA; NU23-05-00095 (Other Grant/Funding Number: AZV, Ministry of Health of the Czech Republic)
Record Dates: First submitted 2023-04-11; First posted 2023-05-16 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Infection; Invasive Pulmonary Aspergillosis
Keywords: biomarkers; qualitative polymerase chain reaction (qPCR); metallomics; mass spectrometry; colonisation; invasive pulmonary aspergillosis; Pentraxin-3
MeSH Terms: conditions — Respiratory Tract Infections; Invasive Pulmonary Aspergillosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — BALF and/or ETA and serum, tissue biopsy (if available), urine (in intubated patients)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspicion of IPA at enrolment: Study subjects with suspicion of IPA at enrolment will be included in this study group.
  Interventions: Diagnostic Test: Next generation improvement of early invasive aspergillosis
- Probable or proven IPA at enrolment: Study subjects with probable or proven IPA at enrolment will be included in this study group.
  Interventions: Diagnostic Test: Next generation improvement of early invasive aspergillosis

INTERVENTIONS:
Diagnostic Test: Next generation improvement of early invasive aspergillosis — Next generation improvement of early invasive aspergillosis test is intended to determine the suitability of new potential biomarkers of aspergillosis.

SUMMARY:
The last decade has seen a significant increase in secondary Aspergillus infections, not only due to primary hypersensitivity, and immunodeficiency based on oncological diseases and their therapy, but mainly due to a rise in severe respiratory infections (H1N1, COVID-19, bacterial infections). This is most evident in critically ill patients whose life is threatened by invasive pulmonary aspergillosis (IPA), with over 90 % of cases being caused by Aspergillus fumigatus. In recent decades, various biomarkers with well-known limits of use (Aspergillus DNA, galactomannan, 1,3-ß-D-glucan) have been used for early diagnosis of IPA. However, the clinical need to clearly distinguish the onset of IPA from colonization is much more significant. The current biomarkers only provide "probable IPA" interpretation, and the diagnosis is rarely confirmed. Based on our preliminary studies, the use of new low molecular weight substances (secondary metabolites) combined with acute-phase proteins (pentraxin 3) allows very reliable immediate confirmation of IPA. In tissue samples, bronchoalveolar lavage fluid, endotracheal aspirate, breath condensate, serum, and urine of critically ill patients, the investigators will be able to recognize and confirm IPA in time using highly sensitive mass spectrometry detecting specific microbial siderophores in correlation with a significantly increased concentration of acute-phase host protein (pentraxin 3) within hours of the beginning of the invasion of lung tissue. Through a prospective multicentre study, the investigators will evaluate the benefit of new biomarkers in non-invasive IPA confirmation, improve the IPA diagnostic algorithm and transfer the detection method to MALDI-TOF spectrometers widely used in Clinical laboratories in the Czech Republic. In MALDI-TOF mass spectrometry, the ion source is matrix-assisted laser desorption/ionization (MALDI), and the mass analyser is a time-of-flight (TOF) analyser.

The study results will contribute to a high clarity of IPA cases, the accurate introduction of antifungal therapy, and a better prognosis of survival of critically ill patients.

DETAILED DESCRIPTION:
This is a prospective study of threshold-driven and continuous response variables from independent control and experimental groups of subjects. The intensive care units in the five hospitals include 63 beds and will provide 2292 potentially suitable critically ill subjects annually during a 3-year prospective study.

In patients with suspected IPA, all types of samples will be collected twice a week for analysis from the date of diagnosis until at least 2 consecutive negative results are obtained, or the patient will be discharged from an intensive care unit. If available, stored aliquots of samples taken 14 - 1 days before the day of diagnosis (mainly the serum and BALF/ETA (bronchoalveolar lavage fluid/endotracheal aspirate) used for galactomannan screening) will be used for Pentraxin 3 (PTX3), Aspergillus qPCR, and HPLC-ESI-FTICR analyses. Results will be reported to clinicians in variable time frames depending on the centre.

The control and experimental group sizes are expected to be approximately equal. Based on the previous experimental and published data, the expected AUC value is 0.8 for the power of study limiting laboratory assay. For Ptx3 and qPCR Aspergillus, a sample size of 13 in each group will be sufficient to detect a significant difference, assuming a power of 80%, and a two-sided significance level of 0.05. The second assay used in the study would require only 7 subjects in each group based on a mean difference of 4303 and an estimated standard deviation of 2500 to detect significant differences assuming the power of 80%, a two-sided significance level of 0.05, and the t-test. When an appropriate threshold is applied to the latter assay, the expected AUC value is 0.99, thus rendering the minimum required number of subjects to 3 for each study group. The investigators expect to enrol more subjects (up to a total of 90) to allow for a possible variation of the values in the groups. Statistical analysis for clinical samples will be performed in R 4.0.2 using standard libraries for exploratory data analysis. Descriptive statistics will be reported in the form of mean, median, standard deviation, standard error of the mean, and coefficient of variation. Differences in male proportion and age will be evaluated using the Wilcoxon rank-sum test for equal variance. Sample frequency will be compared with Fisher's exact test. The normal distribution of the data (age and gender) will be tested using the Shapiro-Wilk normality test. If the data do not meet the normality requirement, the nonparametric Kruskal-Wallis test will be followed by the post hoc pairwise Wilcoxon signed-rank test for further data analysis; for all above-mentioned tests, p <0.05 will be considered statistically significant. R library cutpointr estimates the optimal cut-off value, and the ROC characteristics, specificity, and sensitivity will be determined. Maximize spline, gam, and loss estimates for metrics accuracy and a sum of sensitivity and specificity, and Kernel estimate for Youden index methods will be used for cut-off value estimates. False-negative and false-positive rates will be calculated as controls based on probable IPA and non-IPA.

Patients with suspected IPA defined by the presence of host factors, suggestive imaging, and clinical symptoms, according to the 2008 consensus definitions from the European Organization for the Research and Treatment of Cancer / Mycoses Study Group Education and Research Consortium (EORTC/MSGERC) revised in 2019, will be prospectively recruited in five hospital centres in the Czech Republic from 1st June 2023 to 31st December 2025 (Cohort 1). Mycological and clinical investigations will be performed according to the usual procedures in each centre (imaging, mycological culture, identification using microscopy, and histopathological examination). Molecular detection of hyphae recognized in tissue samples, BALF, and/or ETA will be performed using Aspergillus quantitative PCR (qPCR). IPA-specific acute phase biomarker PTX3 elevation will be analysed in BALF and/or ETA and serum commercial PTX3 immunoassays. Mass spectrometry identification of specific Aspergillus siderophores TafC, TafB, Fc, and secondary metabolite Gtx in the tissue biopsies (if available), urine, BC (intubated patient), BALF, and/or ETA will be performed using HPLC/ESI-FTICR (co-PI 1). All other investigations and treatments, including treatment for aspergillosis, will be based on the standards of each co-applicant team in accordance with the procedures defined in each centre. Population characteristics, clinical and biological data, underlying conditions, medical history, biology, imaging, time to diagnosis, and treatment will be collected for each patient after enrolment and recorded in each centre using an online Castor EDC (Castor's Decentralized Clinical Trials Platform, www.castoredc.com). Routine detection of galactomannan antigen, 1,3-β-D-glucan, PTX3, and Aspergillus qPCR assay will be performed in accordance with the procedures defined in co-participant Public Health Institute Ostrava and Faculty of Medicine, University of Ostrava. The HPLC/ESI-FTICR analysis will be performed by the Institute of Microbiology, Academy of Sciences of the Czech Republic in Prague. TafC enrichment by affinity purification column will be performed by co-applicant University Hospital Olomouc, and MS analyses (HPLC/ESI-FTICR, ESI-FTICR, and MALDI-TOF) will be performed by co-applicant Institute of Microbiology, Academy of Sciences, Czech Republic in Prague. The day of sampling of the first histological or positive mycological specimen will be defined as day 0 (D0). Patients will be classified at month 6 as having a possible, probable, or proven IPA according to the 2019 EORTC/MSGERC criteria.

ELIGIBILITY:
Inclusion Criteria:

* respiratory rate ≥ 30 breaths/min
* PaO2/FiO2 ratio ≤ 250
* multilobar infiltrates
* confusion/disorientation
* uremia (blood urea nitrogen level ≥ 20mg/dL)
* leucocytosis (white blood cell count > 12000/mL) or
* leukopenia (white blood cell count < 4 x 109/L)
* thrombocytopenia (platelet count < 100 x 109/L)
* hyperthermia (core temperature > 38 °C)
* hypothermia (core temperature < 36 °C)
* hypotension requiring aggressive fluid resuscitation
* invasive mechanical ventilation and septic shock requiring vasopressors
* Bronchoalveolar Lavage Fluid (BALF) and/or Endotracheal Aspirate (ETA)

Exclusion Criteria:

- patients, in whom PTX3, Aspergillus qPCR, and HPLC-FTICR were not performed or were performed after the start of antifungal treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients (>18 years) with any respiratory symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of IPA on mass spectrometry | 31 months
  IPA in time will be recognized and analysed in tissue samples (bronchoalveolar lavage fluid, endotracheal aspirate, breath condensate, serum, and urine) of critically ill patients using highly sensitive mass spectrometry detecting specific microbial siderophores in correlation with a significantly increased concentration of acute-phase host protein (pentraxin 3) within hours of the beginning of the invasion of lung tissue. The study results will contribute to a high clarity of IPA cases, the accurate introduction of antifungal therapy, and a better prognosis of survival of critically ill patients in a prospective study of threshold driven and a continuous response variable from independent control and experimental groups of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Jozef Škarda, Assoc.Prof.,MD,DVM,PhD, Principal Investigator — University Hospital Ostrava
Locations (7):
- Czechia (7):
  - Havířov Hospital, Havířov, Moravian-Silesian Region
  - Krnov Hospital, Krnov, Moravian-Silesian Region
  - Public Health Institute Ostrava, Ostrava, Moravian-Silesian Region
  - University of Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - Municipal Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Olomouc, Olomouc, Olomouc Region

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

REFERENCES:
- [Background] Latge JP, Chamilos G. Aspergillus fumigatus and Aspergillosis in 2019. Clin Microbiol Rev. 2019 Nov 13;33(1):e00140-18. doi: 10.1128/CMR.00140-18. Print 2019 Dec 18. PMID 31722890
- [Background] Dobias R, Jaworska P, Tomaskova H, Kanova M, Lyskova P, Vrba Z, Holub C, Svobodova L, Hamal P, Raska M. Diagnostic value of serum galactomannan, (1,3)-beta-d-glucan, and Aspergillus fumigatus-specific IgA and IgG assays for invasive pulmonary aspergillosis in non-neutropenic patients. Mycoses. 2018 Aug;61(8):576-586. doi: 10.1111/myc.12765. Epub 2018 Jun 11. PMID 29575150
- [Background] Koehler P, Bassetti M, Chakrabarti A, Chen SCA, Colombo AL, Hoenigl M, Klimko N, Lass-Florl C, Oladele RO, Vinh DC, Zhu LP, Boll B, Bruggemann R, Gangneux JP, Perfect JR, Patterson TF, Persigehl T, Meis JF, Ostrosky-Zeichner L, White PL, Verweij PE, Cornely OA; European Confederation of Medical Mycology; International Society for Human Animal Mycology; Asia Fungal Working Group; INFOCUS LATAM/ISHAM Working Group; ISHAM Pan Africa Mycology Working Group; European Society for Clinical Microbiology; Infectious Diseases Fungal Infection Study Group; ESCMID Study Group for Infections in Critically Ill Patients; Interregional Association of Clinical Microbiology and Antimicrobial Chemotherapy; Medical Mycology Society of Nigeria; Medical Mycology Society of China Medicine Education Association; Infectious Diseases Working Party of the German Society for Haematology and Medical Oncology; Association of Medical Microbiology; Infectious Disease Canada. Defining and managing COVID-19-associated pulmonary aspergillosis: the 2020 ECMM/ISHAM consensus criteria for research and clinical guidance. Lancet Infect Dis. 2021 Jun;21(6):e149-e162. doi: 10.1016/S1473-3099(20)30847-1. Epub 2020 Dec 14. PMID 33333012
- [Background] Pfister J, Summer D, Petrik M, Khoylou M, Lichius A, Kaeopookum P, Kochinke L, Orasch T, Haas H, Decristoforo C. Hybrid Imaging of Aspergillus fumigatus Pulmonary Infection with Fluorescent, 68Ga-Labelled Siderophores. Biomolecules. 2020 Jan 22;10(2):168. doi: 10.3390/biom10020168. PMID 31979017
- [Background] Alanio A, Delliere S, Fodil S, Bretagne S, Megarbane B. Prevalence of putative invasive pulmonary aspergillosis in critically ill patients with COVID-19. Lancet Respir Med. 2020 Jun;8(6):e48-e49. doi: 10.1016/S2213-2600(20)30237-X. Epub 2020 May 20. No abstract available. PMID 32445626
- [Background] Henneberg S, Hasenberg A, Maurer A, Neumann F, Bornemann L, Gonzalez-Menendez I, Kraus A, Hasenberg M, Thornton CR, Pichler BJ, Gunzer M, Beziere N. Antibody-guided in vivo imaging of Aspergillus fumigatus lung infections during antifungal azole treatment. Nat Commun. 2021 Mar 17;12(1):1707. doi: 10.1038/s41467-021-21965-z. PMID 33731708
- [Background] Meersseman W, Lagrou K, Maertens J, Wilmer A, Hermans G, Vanderschueren S, Spriet I, Verbeken E, Van Wijngaerden E. Galactomannan in bronchoalveolar lavage fluid: a tool for diagnosing aspergillosis in intensive care unit patients. Am J Respir Crit Care Med. 2008 Jan 1;177(1):27-34. doi: 10.1164/rccm.200704-606OC. Epub 2007 Sep 20. PMID 17885264
- [Background] Cao XJ, Li YP, Xie LM, Zhang HL, Qin YS, Guo XG. Diagnostic Accuracy of Bronchoalveolar Lavage Fluid Galactomannan for Invasive Aspergillosis. Biomed Res Int. 2020 Nov 30;2020:5434589. doi: 10.1155/2020/5434589. eCollection 2020. PMID 33335924
- [Background] Khan A, Singh P, Srivastava A. Synthesis, nature and utility of universal iron chelator - Siderophore: A review. Microbiol Res. 2018 Jul-Aug;212-213:103-111. doi: 10.1016/j.micres.2017.10.012. Epub 2017 Nov 2. PMID 29103733
- [Background] Schrettl M, Bignell E, Kragl C, Sabiha Y, Loss O, Eisendle M, Wallner A, Arst HN Jr, Haynes K, Haas H. Distinct roles for intra- and extracellular siderophores during Aspergillus fumigatus infection. PLoS Pathog. 2007 Sep 28;3(9):1195-207. doi: 10.1371/journal.ppat.0030128. PMID 17845073
- [Background] Skriba A, Pluhacek T, Palyzova A, Novy Z, Lemr K, Hajduch M, Petrik M, Havlicek V. Early and Non-invasive Diagnosis of Aspergillosis Revealed by Infection Kinetics Monitored in a Rat Model. Front Microbiol. 2018 Oct 8;9:2356. doi: 10.3389/fmicb.2018.02356. eCollection 2018. PMID 30349512
- [Background] Luptakova D, Pluhacek T, Petrik M, Novak J, Palyzova A, Sokolova L, Skriba A, Sediva B, Lemr K, Havlicek V. Non-invasive and invasive diagnoses of aspergillosis in a rat model by mass spectrometry. Sci Rep. 2017 Nov 28;7(1):16523. doi: 10.1038/s41598-017-16648-z. PMID 29184111
- [Background] Pluhacek T, Lemr K, Ghosh D, Milde D, Novak J, Havlicek V. Characterization of microbial siderophores by mass spectrometry. Mass Spectrom Rev. 2016 Jan-Feb;35(1):35-47. doi: 10.1002/mas.21461. Epub 2015 May 15. PMID 25980644
- [Background] Kamei K, Watanabe A. Aspergillus mycotoxins and their effect on the host. Med Mycol. 2005 May;43 Suppl 1:S95-9. doi: 10.1080/13693780500051547. PMID 16110799
- [Background] Raffa N, Keller NP. A call to arms: Mustering secondary metabolites for success and survival of an opportunistic pathogen. PLoS Pathog. 2019 Apr 4;15(4):e1007606. doi: 10.1371/journal.ppat.1007606. eCollection 2019 Apr. No abstract available. PMID 30947302
- [Background] Vidal-Garcia M, Sanchez-Chueca P, Domingo MP, Ballester C, Roc L, Ferrer I, Revillo MJ, Pardo J, Galvez EM, Rezusta A. Disseminated aspergillosis in an immunocompetent patient with detectable bis(methylthio)gliotoxin and negative galactomannan. Rev Iberoam Micol. 2017 Jan-Mar;34(1):49-52. doi: 10.1016/j.riam.2016.05.007. Epub 2016 Dec 9. PMID 27939578
- [Background] Lehrnbecher T, Hassler A, Groll AH, Bochennek K. Diagnostic Approaches for Invasive Aspergillosis-Specific Considerations in the Pediatric Population. Front Microbiol. 2018 Mar 26;9:518. doi: 10.3389/fmicb.2018.00518. eCollection 2018. PMID 29632518
- [Background] Moura S, Cerqueira L, Almeida A. Invasive pulmonary aspergillosis: current diagnostic methodologies and a new molecular approach. Eur J Clin Microbiol Infect Dis. 2018 Aug;37(8):1393-1403. doi: 10.1007/s10096-018-3251-5. Epub 2018 May 13. PMID 29754210
- [Background] Reichenberger F, Habicht JM, Gratwohl A, Tamm M. Diagnosis and treatment of invasive pulmonary aspergillosis in neutropenic patients. Eur Respir J. 2002 Apr;19(4):743-55. doi: 10.1183/09031936.02.00256102. PMID 11999005
- [Background] Hoenigl M, Orasch T, Faserl K, Prattes J, Loeffler J, Springer J, Gsaller F, Reischies F, Duettmann W, Raggam RB, Lindner H, Haas H. Triacetylfusarinine C: A urine biomarker for diagnosis of invasive aspergillosis. J Infect. 2019 Feb;78(2):150-157. doi: 10.1016/j.jinf.2018.09.006. Epub 2018 Sep 26. PMID 30267801
- [Background] Orasch T, Prattes J, Faserl K, Eigl S, Duttmann W, Lindner H, Haas H, Hoenigl M. Bronchoalveolar lavage triacetylfusarinine C (TAFC) determination for diagnosis of invasive pulmonary aspergillosis in patients with hematological malignancies. J Infect. 2017 Oct;75(4):370-373. doi: 10.1016/j.jinf.2017.05.014. Epub 2017 May 31. No abstract available. PMID 28576596
- [Background] Patil RH, Luptakova D, Havlicek V. Infection metallomics for critical care in the post-COVID era. Mass Spectrom Rev. 2023 Jul-Aug;42(4):1221-1243. doi: 10.1002/mas.21755. Epub 2021 Dec 2. PMID 34854486
- [Background] Dobias R, Skriba A, Pluhacek T, Petrik M, Palyzova A, Kanova M, Cubova E, Houst J, Novak J, Stevens DA, Mitulovic G, Krejci E, Hubacek P, Havlicek V. Noninvasive Combined Diagnosis and Monitoring of Aspergillus and Pseudomonas Infections: Proof of Concept. J Fungi (Basel). 2021 Sep 6;7(9):730. doi: 10.3390/jof7090730. PMID 34575768
- [Background] Kabbani D, Bhaskaran A, Singer LG, Bhimji A, Rotstein C, Keshavjee S, Liles WC, Husain S. Pentraxin 3 levels in bronchoalveolar lavage fluid of lung transplant recipients with invasive aspergillosis. J Heart Lung Transplant. 2017 Sep;36(9):973-979. doi: 10.1016/j.healun.2017.04.007. Epub 2017 Apr 19. PMID 28487045
- [Background] Almeida MA, Almeida-Silva F, Guimaraes AJ, Almeida-Paes R, Zancope-Oliveira RM. The occurrence of histoplasmosis in Brazil: A systematic review. Int J Infect Dis. 2019 Sep;86:147-156. doi: 10.1016/j.ijid.2019.07.009. Epub 2019 Jul 19. PMID 31330326
- [Background] Oide S, Berthiller F, Wiesenberger G, Adam G, Turgeon BG. Individual and combined roles of malonichrome, ferricrocin, and TAFC siderophores in Fusarium graminearum pathogenic and sexual development. Front Microbiol. 2015 Jan 12;5:759. doi: 10.3389/fmicb.2014.00759. eCollection 2014. PMID 25628608
- [Background] Bossuyt PM, Reitsma JB, Bruns DE, Gatsonis CA, Glasziou PP, Irwig L, Lijmer JG, Moher D, Rennie D, de Vet HC, Kressel HY, Rifai N, Golub RM, Altman DG, Hooft L, Korevaar DA, Cohen JF; STARD Group. STARD 2015: an updated list of essential items for reporting diagnostic accuracy studies. BMJ. 2015 Oct 28;351:h5527. doi: 10.1136/bmj.h5527. PMID 26511519
- [Background] Cilloniz C, Torres A, Niederman MS. Management of pneumonia in critically ill patients. BMJ. 2021 Dec 6;375:e065871. doi: 10.1136/bmj-2021-065871. PMID 34872910
- [Background] De Pauw B, Walsh TJ, Donnelly JP, Stevens DA, Edwards JE, Calandra T, Pappas PG, Maertens J, Lortholary O, Kauffman CA, Denning DW, Patterson TF, Maschmeyer G, Bille J, Dismukes WE, Herbrecht R, Hope WW, Kibbler CC, Kullberg BJ, Marr KA, Munoz P, Odds FC, Perfect JR, Restrepo A, Ruhnke M, Segal BH, Sobel JD, Sorrell TC, Viscoli C, Wingard JR, Zaoutis T, Bennett JE; European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group; National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Revised definitions of invasive fungal disease from the European Organization for Research and Treatment of Cancer/Invasive Fungal Infections Cooperative Group and the National Institute of Allergy and Infectious Diseases Mycoses Study Group (EORTC/MSG) Consensus Group. Clin Infect Dis. 2008 Jun 15;46(12):1813-21. doi: 10.1086/588660. PMID 18462102
- [Background] Donnelly JP, Chen SC, Kauffman CA, Steinbach WJ, Baddley JW, Verweij PE, Clancy CJ, Wingard JR, Lockhart SR, Groll AH, Sorrell TC, Bassetti M, Akan H, Alexander BD, Andes D, Azoulay E, Bialek R, Bradsher RW, Bretagne S, Calandra T, Caliendo AM, Castagnola E, Cruciani M, Cuenca-Estrella M, Decker CF, Desai SR, Fisher B, Harrison T, Heussel CP, Jensen HE, Kibbler CC, Kontoyiannis DP, Kullberg BJ, Lagrou K, Lamoth F, Lehrnbecher T, Loeffler J, Lortholary O, Maertens J, Marchetti O, Marr KA, Masur H, Meis JF, Morrisey CO, Nucci M, Ostrosky-Zeichner L, Pagano L, Patterson TF, Perfect JR, Racil Z, Roilides E, Ruhnke M, Prokop CS, Shoham S, Slavin MA, Stevens DA, Thompson GR, Vazquez JA, Viscoli C, Walsh TJ, Warris A, Wheat LJ, White PL, Zaoutis TE, Pappas PG. Revision and Update of the Consensus Definitions of Invasive Fungal Disease From the European Organization for Research and Treatment of Cancer and the Mycoses Study Group Education and Research Consortium. Clin Infect Dis. 2020 Sep 12;71(6):1367-1376. doi: 10.1093/cid/ciz1008. PMID 31802125
- [Background] Dobias R, Jaworska P, Skopelidou V, Strakos J, Visnovska D, Kanova M, Skriba A, Lyskova P, Bartek T, Janickova I, Kozel R, Cwikova L, Vrba Z, Navratil M, Martinek J, Coufalova P, Krejci E, Ulmann V, Raska M, Stevens DA, Havlicek V. Distinguishing Invasive from Chronic Pulmonary Infections: Host Pentraxin 3 and Fungal Siderophores in Bronchoalveolar Lavage Fluids. J Fungi (Basel). 2022 Nov 12;8(11):1194. doi: 10.3390/jof8111194. PMID 36422015
- [Background] Springer J, Held J, Mengoli C, Schlegel PG, Gamon F, Trager J, Kurzai O, Einsele H, Loeffler J, Eyrich M. Diagnostic Performance of (1-->3)-beta-D-Glucan Alone and in Combination with Aspergillus PCR and Galactomannan in Serum of Pediatric Patients after Allogeneic Hematopoietic Stem Cell Transplantation. J Fungi (Basel). 2021 Mar 22;7(3):238. doi: 10.3390/jof7030238. PMID 33810069
- [Background] Springer J, Loeffler J, Heinz W, Schlossnagel H, Lehmann M, Morton O, Rogers TR, Schmitt C, Frosch M, Einsele H, Kurzai O. Pathogen-specific DNA enrichment does not increase sensitivity of PCR for diagnosis of invasive aspergillosis in neutropenic patients. J Clin Microbiol. 2011 Apr;49(4):1267-73. doi: 10.1128/JCM.01679-10. Epub 2010 Dec 29. PMID 21191054
- [Background] Springer J, White PL, Hamilton S, Michel D, Barnes RA, Einsele H, Loffler J. Comparison of Performance Characteristics of Aspergillus PCR in Testing a Range of Blood-Based Samples in Accordance with International Methodological Recommendations. J Clin Microbiol. 2016 Mar;54(3):705-11. doi: 10.1128/JCM.02814-15. Epub 2016 Jan 6. PMID 26739157
- [Background] Morton CO, White PL, Barnes RA, Klingspor L, Cuenca-Estrella M, Lagrou K, Bretagne S, Melchers W, Mengoli C, Caliendo AM, Cogliati M, Debets-Ossenkopp Y, Gorton R, Hagen F, Halliday C, Hamal P, Harvey-Wood K, Jaton K, Johnson G, Kidd S, Lengerova M, Lass-Florl C, Linton C, Millon L, Morrissey CO, Paholcsek M, Talento AF, Ruhnke M, Willinger B, Donnelly JP, Loeffler J; EAPCRI. Determining the analytical specificity of PCR-based assays for the diagnosis of IA: What is Aspergillus? Med Mycol. 2017 Jun 1;55(4):402-413. doi: 10.1093/mmy/myw093. PMID 28339744
- [Background] White PL, Linton CJ, Perry MD, Johnson EM, Barnes RA. The evolution and evaluation of a whole blood polymerase chain reaction assay for the detection of invasive aspergillosis in hematology patients in a routine clinical setting. Clin Infect Dis. 2006 Feb 15;42(4):479-86. doi: 10.1086/499949. Epub 2006 Jan 17. PMID 16421791
- [Background] Lyon GM, Abdul-Ali D, Loeffler J, White PL, Wickes B, Herrera ML, Alexander BD, Baden LR, Clancy C, Denning D, Nguyen MH, Sugrue M, Wheat LJ, Wingard JR, Donnelly JP, Barnes R, Patterson TF, Caliendo AM; AsTeC, IAAM, EAPCRI Investigators. Development and evaluation of a calibrator material for nucleic acid-based assays for diagnosing aspergillosis. J Clin Microbiol. 2013 Jul;51(7):2403-5. doi: 10.1128/JCM.00744-13. Epub 2013 Apr 24. PMID 23616459
- [Background] Thiele C, Hirschfeld G. Confidence intervals and sample size planning for optimal cutpoints. PLoS One. 2023 Jan 3;18(1):e0279693. doi: 10.1371/journal.pone.0279693. eCollection 2023. PMID 36595525